CLINICAL TRIAL: NCT04540484
Title: The Prevalence of SARS-CoV-2 IgG Antibody Formation in Physicians at Advocate Lutheran General Hospital and Their Household Members
Brief Title: COVID-19 IgG Formation in Physicians at ALGH and Their Household Members
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 1606472-1; M5500436 (Other: ALGH)
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2022-02

CONDITIONS: Covid19; SARS-CoV Infection; Communicable Disease
Keywords: COVID19; IgG Testing; COVID-19 Antibodies
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Communicable Diseases | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALGH Physicians: Attending physicians on the medical staff, fellow physicians, and resident physicians that work at Advocate Lutheran General Hospital (ALGH) from March 1st, 2020 and forward.
  Interventions: Other: Screening
- Household Members: Household members above age 18 who lived in household of ALGH physician who tested positive for COVID-19 IgG antibodies, and who lived with that physician for at least 2 consecutive weeks.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Blood test screening for covid
  Other Names: Screening for COVID

SUMMARY:
This study is a community hospital-based study that will enhance information being obtained in similar studies taking place in France, Denmark, and China. These studies are designed to assess risk of healthcare workers during outbreaks of Coronavirus 2019 (COVID-19) also known as sudden acute respiratory syndrome-coronavirus-2 (SARS-CoV-2). This will be a prospective, single-center observational study involving human subjects. IgG (Immunoglobulin G) antibody will be tested in the serum of physicians working at Advocate Lutheran General Hospital (ALGH). IgG antibodies are the antibodies that form in response to viral or bacterial infections and typically reflect protection against said infection. To date, there have been no studies confirming that IgG antibody formation confers immunity, but studies are ongoing. Furthermore, data is lacking showing conclusive persistence of (possibly protective) antibodies over time. Attending physicians on the medical staff, fellow physicians, and house staff residents who worked at ALGH from March 1st, 2020 and on, will be eligible for the study. Testing will involve a venipuncture to obtain approximately 3mL of blood to be sent to ACL Laboratories for SARS-CoV-2 IgG testing. For physician subjects, this will be performed on four separate occasions, once at the onset of the study, a second test 3 months after the first test, a third test 6 months from the time of the first test, and a fourth and final test 12 months after the initial test. Two household members (defined below), one-time testing will occur within 2 weeks of the physician subject testing positive. All testing will be performed in a two-week window. All physician subjects will be tested at a centralized site that is only serving these subjects, by appointment. We will be offloading testing for household members to one localized commercial ACL site on the ALGH campus at the Center for Advanced Care. The household member testing will be extended to an additional two-week period after the two week window in which physicians are tested for a total of four weeks maximum. One-time testing for IgG antibodies to COVID-19 will be offered to a maximum of two household members, as defined as, any person over the age of 18 years old who has lived at home with the physician, who has tested positive for IgG antibodies, for at least 2 weeks in total duration since March 1st, 2020. The physician will be permitted to choose who gets tested, and the chosen adult subject will provide their independent consent to be tested.

DETAILED DESCRIPTION:
Study is complete. Data analysis is being put together.

ELIGIBILITY:
Inclusion Criteria:

* Attending physician staff members, fellow physicians, and resident house staff members who were on staff at ALGH from March 1st, 2020 and on, with potential exposure to COVID-19 patients.
* A maximum of two adult household members as defined as, any person over the age of 18 years old who has lived at home with the physician for at least 2 weeks in total duration since March 1st, 2020. Any adult household member of attending physicians on the medical staff, fellow physicians, and resident physicians may qualify as long as the tested physician resulted positive for IgG Antibodies to COVID-19. The adult household member will be selected by the household physician based on their assessment of risk of also testing positive.
* Must be willing to undergo venipuncture, sign consent and complete the questionnaire. Participants need to speak, read, and understand English at the literacy level of a 8th grader.
* Those with a prior documented COVID-19 infection are eligible for study inclusion. We will rely on self-reporting by physicians due to the fact that the data from the other study conducted in the Advocate Aurora System has been de-identified and we cannot access the results on individual participants in our study.

Exclusion Criteria:

* Healthcare providers and/or their household members who would not want venipuncture performed on them
* Healthcare workers who are not on the medical staff or members of the resident house staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advocate Lutheran General Hospital Physicians and their household members.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Identifying positive COVID-19 IgG formation | up to 1 year

SECONDARY OUTCOMES:
Physician Prevalence of COVID-19 serum IgG | up to 1 year
  The prevalence of COVID-19 serum IgG in physician participants at study entry, 3 months, 6 months, and 12 months after enrollment.
Household Member Prevalence of COVID-19 serum IgG | up to 1 year
  The prevalence of COVID-19 serum IgG in household members (as defined above) of physician participants that are positive at the time the associated physician tested positive.
Physician Risk of Exposure | up to 1 year
  The differences in prevalence of COVID-19 IgG in physician participants that are deemed to be at minimum, moderate or high risk of COVID-19 exposure.
Physician and Household Member Transmission | up to 1 year
  The differences in prevalence of COVID-19 IgG in household members of physician participants that are positive for COVID-19 IgG.
Asymptomatic Infection | 1 year
  The correlation between IgG prevalence and previous COVID-19 symptoms - a means of quantifying the presence of asymptomatic carriers amongst the medical staff, an important and heretofore poorly described vector of transmission.
PPE Use and Positivity | up to 1 year
  The correlation between the prevalence of seropositivity and adherence to best practices regarding the use of personal protective equipment.
Antibody Persistence | up to 1 year
  The development of COVID19 infections in physicians at our hospital over the test period of 12 months, and its correlation to Covid19_IgG positivity. This will allow us to understand the persistence of the antibody and its potential neutralizing power, over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No